CLINICAL TRIAL: NCT03080376
Title: Home Exercise Intervention in Childhood Obesity: Randomized Clinical Trial Comparing Print-based Versus Web-based Platform
Brief Title: Home Exercise Intervention in Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine Department, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-5
Record Dates: First submitted 2017-03-05; First posted 2017-03-15 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Child Obesity
Keywords: Exercise; Web-based intervention
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Web-based intervention without support (Experimental): 3 months Web-based intervention without support
  Interventions: Other: Web-based intervention without support
- Web-based intervention with support (Experimental): 3 months Web-based intervention with support (e-mails)
  Interventions: Other: Web-based intervention with support
- Traditional intervention (Active Comparator): 3 months of Printed-based intervention
  Interventions: Other: Traditional intervention

INTERVENTIONS:
Other: Web-based intervention with support — Web-based combined aerobics and muscular strength exercises.
  Arms: Web-based intervention with support
Other: Web-based intervention without support — Web-based combined aerobics and muscular strength exercises.
  Arms: Web-based intervention without support
Other: Traditional intervention — 3 months of Printed-based combined aerobics and muscular strength exercise intervention.
  Arms: Traditional intervention

SUMMARY:
Aim: To evaluate the impact of a physical exercise Web-based program with or without support on body composition, physical fitness and blood pressure values.

Design: Randomized Controlled Trial. Population: Obese children and adolescents.

DETAILED DESCRIPTION:
In recent years there has been a decline in levels of physical activity (PA) in both children and adults. The promotion of PA is also a key element in the treatment of obesity, along with changing eating habits, but usually has very low levels of adherence. Active video games may be an alternative for the promotion of PA in the treatment of obesity.

The objective of this project is to evaluate the impact of a physical exercise Web-based program with or without support on Body Composition, Physical Fitness and Blood Pressure values.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese children and adolescents

Exclusion Criteria:

* Secondary obesity syndromes
* Severe obesity (z score > 2.5)

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of body fat | Change from Baseline Percentage of body fat at 3 months
  Percentage of body fat

SECONDARY OUTCOMES:
Hand strength | Change from Baseline Hand strength at 3 months
  Hand strength
Oxygen consumption peak | Change from Baseline Oxygen consumption peak at 3 months
  Oxygen consumption peak
Blood pressure | Change from Baseline Blood Pressure at 3 months
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: JF Lisón, Dr, Study Director — University CEU Cardenal Herrera
Locations (1):
- Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No